CLINICAL TRIAL: NCT06967792
Title: Evaluation of the Safety of Terahertz Scanning System on Corneas: Phase I Trial
Brief Title: Evaluation of the Safety of Terahertz Scanning System on Corneas
Status: Recruiting | Type: Observational
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: R2022-2604
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Corneal Diseases
Keywords: cornea; corneal edema; Terahertz; hydration
MeSH Terms: conditions — Corneal Diseases; Corneal Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blind group: Eyes that are deemed functionally blind but contain healthy corneas.
  Interventions: Device: Terahertz (THz) scanning using THz Imaging system.

INTERVENTIONS:
Device: Terahertz (THz) scanning using THz Imaging system. — The Terahertz (THz) scanning system is non-invasive and non-contact. It is a prototype developed by Institute of Materials Research and Engineering (IMRE), A*STAR, Singapore and is performed for the purpose of research. THz scanning will provide safety data in human and the measurement of cornea hydration status. Each THz scan will take approximately 1 second. Real-time data will be generated when participants are positioned in front of the device.

SUMMARY:
This observational study aims to establish the safety profile of the use of Terahertz (THz) scanning system on corneal diseases. Participants with "non-seeing" eyes but normal corneas will undergo THz scanning. Eye examinations will be conducted at baseline, immediately after scanning, and at 1 day, 1 week, and 1 month post-scanning. These examinations will include measurements of visual acuity, eye structural, retinal health, corneal cell morphology, and corneal nerve status. The investigators hypothesize that the THz scanning system is safe for application to the human cornea.

DETAILED DESCRIPTION:
Corneal disease is the second leading cause on irreversible blindness in the world. There are more than 250 million people living with visual acuity loss or blindness globally. The cornea is a transparent and avascular tissue that consists of 78% water by volume. With its high-water content, the homogeneity of corneal stromal tissue and the lack of physiological variations allows Terahertz (THz) imaging to be a promising method for sensing corneal hydration level as it is highly sensitive to water. The water content of the cornea is regulated by passive and active mechanism to ensure the preservation of essential transmission and focusing properties. When there is an abnormal elevation of water concentration in the cornea (>5% above the physiological level), it will lead to a significant change in the amount of scattered light and the gradual loss of corneal transparency, this is known as corneal opacification which can be due to corneal edema or corneal scarring. Corneal opacity is one of the leading causes of reversible blindness and visual impairment. When corneal opacity progresses to the end-stage disease, the current and only option would be undergoing corneal transplantation. However, there is a global shortage of donor corneas furthermore, patients who undergo corneal transplantation would require life-long topical immunosuppressant. Hence, monitoring the progression of corneal edema or corneal scarring is essential to help prevent the disease from reaching the end stage. However, a direct marker for the evaluation of corneal edema remains lacking.

THz waves are electromagnetic radiation, and have emerged as a novel, non-invasive and non-contact imaging modality in the biomedical field, with a fast-scanning speed (30ms per scan) to meet medical diagnostic needs. With its fast scanning, it provides a more accurate result for the estimation of corneal thickness. Its high sensitivity hydration absorption and characterization peaks of collagen will provide a useful tool to obtain information that are related to the corneal layers. Water has a high dielectric constant and is highly absorptive to THz spectrum. This allows THz wave to be highly sensitive to water content in tissue. Furthermore, THz scan has been applied to a variety of hydration-related diseases or conditions. With THz scan, early detection of disease and diagnosis can be carried out. Some examples would be the prediction of skin flap failure, diagnosis for the presence of caries lesion at its initial stage, identification of skin cancer in skin biopsy samples and to access the physiological dynamics of tear film in dry eye syndrome. Previous studies have demonstrated that THz scanning system could be used as an early diagnostic tool, to identify the cancerous area based on the lack of clear cellular order in the skin. It was able to detect disease conditions in deeper layers, allowing it to be an effective early diagnostic tool for basal cell carcinoma. Moreover, it had been confirmed that THz scanning system had the sensitivity to identify the difference in colon tissue composition. The findings showed that the properties of ex vivo tissue, had an increase in both absorption coefficient and refractive indices in disease tissue when compared to healthy tissue. A recent study showed that with THz scanning system, clinicians will be able to obtain different images, such as 3D imaging methods to provide multiple views of internal structures. Furthermore, with the THz scan, the process of water loss in an in vitro porcine corneal tissue could be determined using a THz reflection imaging system. It was found that THz wave was approximately linear to the water content concentration, and that the slope decreased monotonously with an increase in frequency. These results suggest that THz imaging can be used for the clinical diagnosis of corneal edema or scars, dry eye diseases and corneal hydration in refractive surgery. With this, investigators would like to conduct this study to ascertain the safety of THz imaging system on humans.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age
* Regardless of gender (Male/Female)
* Regardless of race (Chinese/Malay/Indian/Eurasian/Others)
* Willingness and ability to follow all instructions and comply with study schedule for study visit
* Have at least 1 eye (Study eye) that is deemed functionally blind but contain healthy corneas
* Ability to hold face sufficiently stable to undergo necessary scans
* Best Spectacle Corrected Visual Acuity (BSCVA) in the study eye of hand motion or worse

Exclusion Criteria:

* Pregnant/Breast-feeding women
* Eyes with previous major surgery on the cornea such as corneal transplantation, refractive surgery, corneal cross-linking procedure
* Eyes with previous infectious keratitis
* Eyes with long-term use of glaucoma eye drops
* Eyes with known moderate or server meibomian gland dysfunction
* Eyes with active inflammation or infection, or chronic ocular surface inflammation
* Systemic diseases that affect the ocular surface, such as systemic autoimmune diseases

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 5 participants who have unilateral or bilateral functionally blind eyes with normal corneas will be recruited from Singapore National Eye Centre.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Level of visual acuity | 1 month
  Participants will undergo visual acuity assessment including uncorrected distance visual acuity (UDVA) and corrected distance visual acuity (CDVA) using Snellen chart at every visit. The last line on the chart that subjects are able to read correctly will be selected to calculate the visual acuity.

SECONDARY OUTCOMES:
National Eye Institute (NEI) Score | 1 month
  The cornea will be divided into five regions, each scored ranging from 0 (no fluorescein staining) to 3 (severe fluorescein staining) according to the grading scheme. The total NEI score will range from 0 to 15.
Extent of anterior chamber (AC) inflammation | 1 month
  AC cells will be graded by the Standardization of Uveitis Nomenclature Working Group on the ordinal scale of 0(<1 cell/1 square millimeter, high-intensity beam), 0.5+ (1 to 5 cells/beam), 1+ (6 to 15 cells/beam), 2+ (16 to 25 cells/beam), 3+ (26 to 50 cells/beam), or 4+ (more than 50 cells/beam).
Lens density grade | 1 month
  Lens density will be also evaluated using the Pentacam device. Pentacam Nuclear Staging will provide a cataract grading score on an ordinal scale (from 0 to 5).
Level of anterior chamber (AC) flare | 1 month
  AC flare will be graded on the ordinal scale of 0 (none), 1+ (faint), 2+ (moderate; iris and lens details clear), 3+ (marked; iris and lens details hazy), or 4+ (fibrin or plastic aqueous).
Level of conjunctival hyperemia | 1 month
  The conjunctival hyperemia will be graded by the Food and Drug Administration (FDA) grading scale: 0 (None), 1 (Trace), 2 (Mild), 3 (Moderate), and 4 (Severe).
Severity of lens opacity | 1 month
  The lens opacity will be graded using the Lens Opacities Classification System III (LOCS III).
Central corneal thickness | 1 month
  Central corneal thickness (CCT) will be assessed using Anterior Segment Optical Coherence Tomography. The CCT will be measured using a build-in caliper software.
Corneal endothelium morphology profiles | 1 month
  Specular Microscopy will be used to examine eight morphometric parameters of the corneal endothelium.
Extent of keratocytes activation | 1 month
  In vivo confocal microscopy will be used to capture images of keratocytes. The gray values of reflectivity for corneal stromal scans will be semi-quantified to confirm if there are significant changes in the activity of stromal keratocytes.
Fundus healthy status | 1 month
  The fundus photographs will be taken 30 minutes after instillation of dilation eye drops (1% tropicamide (Alcon, USA) and a detailed evaluation of changes in fundus health will be made by an ophthalmologist.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No